CLINICAL TRIAL: NCT00579371
Title: Cadaveric Islet Transplantation in Patients With Insulin-Dependent Diabetes Mellitus
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per Coordinator: study was closed and no cadaveric implants were performed
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0149-03-XX; BB IND 11397 (Other: FDA)
Record Dates: First submitted 2007-12-17; First posted 2007-12-24 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Islets of Langerhans Transplantation; Diabetes Mellitus, Type 1
Keywords: islet transplantation; type 1 diabetes mellitus; steroid-free immunosuppression; rabbit anti-thymocyte globulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Transplantation of Islets of Langerhans (Experimental): Subjects will receive islets isolated from one donor pancreas per transplantation event. Subjects will receive a cumulative dose of 8,000 International Units/kg. Islets will be infused intraportally. If necessary, additional transplantation events will be performed.
  Interventions: Drug: Islets of Langerhans

INTERVENTIONS:
Drug: Islets of Langerhans — Subjects will receive islets isolated from one donor pancreas per transplantation event. Subjects will receive a cumulative dose of 8,000IE/kg. Islets will be infused intraportally. If necessary, additional transplantation events will be performed.
  Other Names: transplanted islets of Langerhans

SUMMARY:
We hypothesize that the following improvements to islet transplantation will increase the islet mass successfully isolated and allow for engraftment from a single pancreas. The improvements are:

* Using Two-Layer method preservation to improve pancreas quality before islet isolation
* Maintaining isolated islets in culture before transplantation
* Using a steroid-free immunosuppression regimen
* Transplanting the best combination of donor and recipient possible after human leukocyte antigens (HLA) screening and final crossmatching

DETAILED DESCRIPTION:
We hypothesize that the following improvements to islet transplantation will increase the islet mass successfully isolated and allow for engraftment from a single pancreas:

using Two-Layer method preservation to improve pancreas quality before islet isolation, maintaining isolated islets in culture before transplantation, using a steroid-free immunosuppression regimen, and transplanting the best combination of donor and recipient possible after HLA screening and final crossmatching.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Diagnosis of Type-1 diabetes mellitus for more than 5 years with at least one of the following complications:

  * Metabolic lability/instability (two or more episodes of severe hypoglycemia) or two or more hospital visits for diabetic ketoacidosis during the previous year
  * Progression of secondary complications of diabetes as determined by The Nebraska Medical Center/University of Nebraska Medical Center staff endocrinologists
* Group 2: Diagnosis of Type-1 diabetes with successful renal transplant on steroid-free, FK506/rapamycin-based immunosuppression

Exclusion Criteria:

* Severe co-existing cardiac disease
* Active alcohol or substance abuse, including cigarette smoking
* Psychiatric disorder making the subject not a suitable candidate for transplantation
* History of medical non-compliance
* Active infection, including hepatitis C and B, HIV, and tuberculosis (or suspected tuberculosis)
* Any history of malignancy except squamous or basal cell skin cancer
* BMI >28 kg/meter-squared, or body weight >80kg at screening visit, or >85kg on the day of transplantation (due to the difficulty of obtaining a sufficiently large islet mass to adequately treat either large patients or those whose obesity elevates their insulin needs)
* Positive C-peptide response to intravenous glucose tolerance test and Mixed Meal glucose tolerance test: any C-peptide >0.3 ng/mL post infusion
* Inability to provide informed consent
* Age less than 19 or greater than 70 years
* Creatinine clearance <60 mL/min/1.73 meter-squared for Group 1 and creatinine clearance <40 mL/min/1.73 meter-squared for Group 2 (those subjects currently on immunosuppression due to previous kidney transplant)
* Macroalbuminuria (urinary albumin excretion rate >300 mg/24h) for Group 1 and macroalbuminuria (urinary albumin excretion rate >600mg/24h) for Group 2
* Baseline Hb <10 gm/dL
* Baseline liver function tests outside of normal range
* Presence of gallstones or hemangioma in liver on baseline ultrasound exam
* Positive pregnancy test, intention of future pregnancy, or presently breast-feeding
* Evidence of sensitization on panel reactive antibodies (PRA)
* Insulin requirement >0.7 IU/kg/day or HbA1c >15%
* Hyperlipidemia
* Under treatment for a medical condition requiring chronic use of steroids
* Use of Coumadin or other anticoagulant therapy (except aspirin) or a prothrombin time/international normalized ratio (PT-INR) >1.5
* Diagnosis of Addison's disease

Additional Exclusion Criteria for Group 2 Subjects:

* Any history of organ transplantation other than kidney or pancreas
* Any previous graft lost to rejection
* Any history of early, multiple, or vascular renal allograft rejection

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-03-17 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Incidence of insulin independence with a single islet transplant | 1 year post-transplantation
  Incidence of insulin independence with a single transplantation measured at one year post-transplantation.

SECONDARY OUTCOMES:
Islet mass resulting in insulin independence/reduced exogenous insulin requirement | 1 year post-transplantation
  Insulin independence or reduced exogenous insulin required measured at one year post-transplantation.
Graft survival | 3 years post-transplantation
  The survival of the Islets of Langerhans graft as measured at three years post-transplantation.
Metabolic functional assessments of the islet graft | 3 years post-transplantation
  An assessment of the metabolic function of the islet of Langerhans graft as measured three years post-transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: R Brian Stevens, MD PhD, Principal Investigator — University of Nebraska
Locations (1):
- The Nebraska Medical Center, Omaha, Nebraska, United States